CLINICAL TRIAL: NCT03370770
Title: GioTag: Real-world Data Study on Sequential Therapy With Gi(l)Otrif®/ Afatinib as First-line Treatment Followed by Osimertinib in Patients With EGFR Mutation Positive Advanced Non-small Cell Lung Cancer
Brief Title: Afatinib Osimertinib Sequencing NIS
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200-0286
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with EGFR mutation-positive NSCLC: (Non-Small Cell Lung Cancer) (Epidermal Growth Factor Receptor)
  Interventions: Drug: Afatinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Afatinib — GILOTRIF, GIOTRIF, XOVOLTIB
Drug: Osimertinib — on T790M resistance mutation was developed

SUMMARY:
This is a non-interventional, multi-country, multi-centre cohort study based on existing data from medical records of patients with EGFR mutation-positive advanced NSCLC treated with afatinib (Gi(l)otrif®) as the first-line treatment followed by osimertinib in case the T790M resistance mutation was developed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with EGFR mutation-positive advanced non-small cell lung cancer (NSCLC)
* The tumour harbours common EGFR mutations (Del19, L858R) at start of first-line treatment
* Patients who initiated second-line osimertinib treatment for acquired T790M mutation at least 10 months prior to data entry, AND who were treated with afatinib (Gi(l)otrif®) in the first-line
* Patients treated with osimertinib within an EAP/CUP or regular clinical practice
* Age ≥ 18 years
* Signed and dated written informed consent per regulations (Exemption of a written informed consent for NIS based on existing data in countries per local regulations and legal requirements)

Exclusion Criteria:

* Patients who received drug(s) other than osimertinib as the second-line treatment and/or patients who received drug(s) other than afatinib (Gi(l)otrif®) as the first-line treatment
* Patients with active brain metastases at start of treatment (either afatinib/Gi(l)otrif® or osimertinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study is planned that around 65 study centres in 11 countries will be participating in this noninterventional study and at least 190 consecutive eligible patients will be enrolled to the study. Every patient who fulfils inclusion and exclusion criteria and agree to participate in the study (if a written informed consent is required for this NIS by local regulation and legal requirement) will be selected until the required sample size is achieved.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Otto-Wagner Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hochmair MJ, Morabito A, Hao D, Yang CT, Soo RA, Yang JC, Gucalp R, Halmos B, Marten A, Cufer T. Sequential afatinib and osimertinib in patients with EGFR mutation-positive non-small-cell lung cancer: final analysis of the GioTag study. Future Oncol. 2020 Dec;16(34):2799-2808. doi: 10.2217/fon-2020-0740. Epub 2020 Aug 28. PMID 32854536
- [Derived] Feinberg B, Halmos B, Gucalp R, Tang W, Moehring B, Hochmair MJ. Making the case for EGFR TKI sequencing in EGFR mutation-positive NSCLC: a GioTag study US patient analysis. Future Oncol. 2020 Aug;16(22):1585-1595. doi: 10.2217/fon-2020-0188. Epub 2020 Aug 6. PMID 32757853
- [Derived] Yamamoto N, Mera T, Marten A, Hochmair MJ. Observational Study of Sequential Afatinib and Osimertinib in EGFR Mutation-Positive NSCLC: Patients Treated with a 40-mg Starting Dose of Afatinib. Adv Ther. 2020 Feb;37(2):759-769. doi: 10.1007/s12325-019-01187-y. Epub 2019 Dec 20. PMID 31863283
- [Derived] Hochmair MJ, Morabito A, Hao D, Yang CT, Soo RA, Yang JC, Gucalp R, Halmos B, Wang L, Marten A, Cufer T. Sequential afatinib and osimertinib in patients with EGFR mutation-positive non-small-cell lung cancer: updated analysis of the observational GioTag study. Future Oncol. 2019 Sep;15(25):2905-2914. doi: 10.2217/fon-2019-0346. Epub 2019 Aug 2. PMID 31370698
- [Derived] Hochmair MJ, Morabito A, Hao D, Yang CT, Soo RA, Yang JC, Gucalp R, Halmos B, Wang L, Golembesky A, Marten A, Cufer T. Sequential treatment with afatinib and osimertinib in patients with EGFR mutation-positive non-small-cell lung cancer: an observational study. Future Oncol. 2018 Nov;14(27):2861-2874. doi: 10.2217/fon-2018-0711. Epub 2018 Oct 19. PMID 30336693
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Non-interventional, multi-centre cohort study based on existing data from medical records of patients with epidermal growth factor receptor (EGFR) mutation-positive advanced non-small cell lung cancer (NSCLC) treated with afatinib (Gi[l]otrif®) as first-line treatment followed by osimertinib in case the T790M resistance mutation was developed. The study included an extension analysis using additional collected data of the enrolled patients.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Only patients that met all the inclusion and none of the exclusion criteria were included in the trial.
Groups:
- Patients With EGFR Mutation-positive NSCLC: Patients with EGFR mutation-positive NSCLC with acquired T790M mutation at least 10 months prior to data entry, and who were treated with afatinib (Gi[l]otrif®) (50mg or 40mg or 30mg or 20mg tablet once daily as indicated in the approved labels of afatinib (Gi[l]otrif®)) in the first-line line treatment followed by second-line osimertinib treatment (80 milligram (mg) or 40 mg tablets once daily as indicated in the approved labels of osimertinib).
Period: Overall Study
Arm/Group | Patients With EGFR Mutation-positive NSCLC
Started | 204
Completed | 98
Not Completed | 106
Not completed — Patient was followed in another hospital center | 1
Not completed — Progressive Disease | 98
Not completed — Adverse Event | 2
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): FAS included all patients who were enrolled into the study, met all inclusion criteria and did not meet any exclusion criteria and provided a written and signed informed consent (if a written informed consent was required for this NIS by local regulation and legal requirement).
Arm/Group | Patients With EGFR Mutation-positive NSCLC
Number analyzed (Participants) | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 181
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 50
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 18
  White | 120
  More than one race | 0
  Unknown or Not Reported | 13

OUTCOME MEASURES:

1. Primary Outcome: Time on Treatment With Afatinib (Gi(l)Otrif®) Followed by Osimertinib
Description: Time on treatment, which was defined as time in months from the start date of Afatinib (Gi[l]otrif®) treatment ('start date of initial dose' for First-Line Treatment) to the end date of Osimertinib treatment (maximum between 'end date of initial dose' and the last 'end date of dose modification' for Second-Line Treatment) or death date due to any cause ('date of death').
  Time on treatment (months) = Time on treatment (days)/30.4375.
  'Time on treatment was analysed using Kaplan-Meier method, and the median along with two-sided 90% confidence interval was displayed using the Greenwood's formula for estimation of standard errors.
Time Frame: Data collected from start of treatment until data entry completion, up to 96.8 months for first analysis and up to 114.1 months for the extension analysis.
Population: Full Analysis Set (FAS): All patients who were enrolled into the study, met all inclusion criteria and did not meet any exclusion criteria and provided a written and signed informed consent. 1 Patient was excluded from extension analysis due to conflicting data on the discontinuation date of osimertinib treatment.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Patients With EGFR Mutation-positive NSCLC
Number analyzed (Participants) | 204
Months
  First analysis | 27.6 [25.9 to 31.3]
  Extension analysis: number analyzed (Participants) | 203
  Extension analysis | 27.7 [26.7 to 29.9]

2. Secondary Outcome: The Percentage of Participants With Different Types of Mutations After Categorisation
Description: Different types of resistance mutations identified at the time of discontinuation of osimertinib treatment were systematically reviewed and categorised.
Time Frame: Data collected from start of treatment until data entry completion; up to 96.8 months.
Population: Patients in the Full Analysis Set (FAS), who discontinued treatment and with positive test results (either EGFR sensitizing Mutation and/or T790M) available.
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Patients With EGFR Mutation-positive NSCLC
Number analyzed (Participants) | 39
Percentage of participants (%)
  T790M positive | 69.2
  Loss of T790M | 20.5
  T790M positive, loss of sensitizing mutation | 10.3

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study, as data were collected retrospectively. The approach was changed for the extension period: Adverse Events were collected from start of data collection once informed consent was signed onwards until the end of data collection, up to 18 months.
Description: Participants in the Full Analysis Set (FAS), who were included in the extension period.
Arm/Group | Patients With EGFR Mutation-positive NSCLC
All-Cause Mortality (participants affected / at risk) | 31/203
Serious Adverse Events (participants affected / at risk) | 32/203
Other Adverse Events (participants affected / at risk) | 62/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With EGFR Mutation-positive NSCLC (N=203)
Disease progression (General disorders) | 27
Death (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With EGFR Mutation-positive NSCLC (N=203)
Diarrhoea (Gastrointestinal disorders) | 52
Stomatitis (Gastrointestinal disorders) | 21
Rash (Skin and subcutaneous tissue disorders) | 34
Dermatitis (Skin and subcutaneous tissue disorders) | 12
Paronychia (Infections and infestations) | 25

LIMITATIONS AND CAVEATS:
This study has no comparator group limiting the interpretability of the results as they cannot be put into perspective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT03370770/SAP_000.pdf
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03370770/Prot_001.pdf